CLINICAL TRIAL: NCT02124395
Title: Assessment of Health-related Quality of Life in Rare Kidney Stone Formers in the Rare Kidney Stone Consortium
Brief Title: Health-related Quality of Life in Rare Kidney Stone
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 13-00968; 1U54DK083908-01 (NIH)
Record Dates: First submitted 2014-04-23; First posted 2014-04-28 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Primary Hyperoxaluria; Cystinuria; Adenine Phosphoribosyl Transferase Deficiency; Dent Disease
MeSH Terms: conditions — Hyperoxaluria, Primary; Cystinuria; Adenine phosphoribosyltransferase deficiency; Dent Disease | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Primary Hyperoxaluria: All rare kidney stone patients enrolled in RKSC registries that are able to communicate using the English language, are able to consent to participation in the study, have internet access with an email account and/or a valid address and are at minimum 5 years of age (for SF-10)
  Interventions: Other: Health-related Quality of Life in Rare Kidney Stone Questionnaire
- Cystinuria: All rare kidney stone patients enrolled in RKSC registries that are able to communicate using the English language, are able to consent to participation in the study, have internet access with an email account and/or a valid address and are at minimum 5 years of age (for SF-10)
  Interventions: Other: Health-related Quality of Life in Rare Kidney Stone Questionnaire
- Dent Disease: All rare kidney stone patients enrolled in RKSC registries that are able to communicate using the English language, are able to consent to participation in the study, have internet access with an email account and/or a valid address and are at minimum 5 years of age (for SF-10)
  Interventions: Other: Health-related Quality of Life in Rare Kidney Stone Questionnaire
- APRT deficiency: All rare kidney stone patients enrolled in RKSC registries that are able to communicate using the English language, are able to consent to participation in the study, have internet access with an email account and/or a valid address and are at minimum 5 years of age (for SF-10)
  Interventions: Other: Health-related Quality of Life in Rare Kidney Stone Questionnaire

INTERVENTIONS:
Other: Health-related Quality of Life in Rare Kidney Stone Questionnaire

SUMMARY:
Assessment of Health-related Quality of Life in Rare Kidney Stone Formers in the Rare Kidney Stone Consortium

DETAILED DESCRIPTION:
The purpose of this study is to learn about Health-related Quality Of Life (HRQoL) in patients enrolled in the Rare Kidney Stone Consortium (RKSC) registries. Quality of life studies look at different aspects of both physical and mental components of people's lives. HRQoL data for people affected by kidney stones are not currently available for people followed over time.

ELIGIBILITY:
Inclusion Criteria:

* Qualify to participate in one of the Rare Kidney Stone Registries.
* Be at least 5 years old (for SF-10)
* Are able to communicate using the English language
* Consent to participate in the study (or "assent" if under 18 years old)
* Have internet access with an email account or a valid home address

Exclusion Criteria:

None, if inclusion criteria are met

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sample will be selected from the Rare Kidney Stone Consortium registries
Sampling Method: Non-Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Assessment of HRQoL in patients with rare kidney stones | Once a year for up to 5 years after signed consent
  Assessment of HRQoL in patients with rare kidney stones. Comparison of HRQoL results between rare kidney stone formers, general population and other populations with relevant chronic diseases

CONTACTS AND LOCATIONS:
Overall Officials: David Goldfarb, MD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (2):
  - Primary Hyperoxaluria and Dent Disease Registry - Mayo Clinic, Rochester, Minnesota
  - New York University School of Medicine - Cystinuria Registry, New York, New York
- APRT Registry - Landspitali Universtiy Hospital, Reykjavik, Iceland

REFERENCES:
- [Background] Modersitzki F, Pizzi L, Grasso M, Goldfarb DS. Health-related quality of life (HRQoL) in cystine compared with non-cystine stone formers. Urolithiasis. 2014 Feb;42(1):53-60. doi: 10.1007/s00240-013-0621-4. Epub 2013 Nov 20. PMID 24253538